CLINICAL TRIAL: NCT04531098
Title: A Bridging Study: Comparing Two Sci-B-Vac™ Batches in Healthy Adults
Brief Title: A Bridging Study: Comparing Two Lots of Sci-B-Vac™ and Engerix-B in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VBI Vaccines Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SG-005-05
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Results first posted 2022-06-24 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Hepatitis B
Keywords: Sci-B-Vac; Prophylactic vaccine; Hepatitis B vaccines; Phase 3; pre-S1; pre-S2; Surface antigen; 3-antigen
MeSH Terms: conditions — Hepatitis B | interventions — Pre-S vaccine; Engerix-B

STUDY DESIGN:
Intervention Model Description: Single blind, three-arm, two-stage, randomized study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sci-B-Vac-SciGen (Experimental): The 3-antigen HepB vaccine, Sci-B-Vac-SciGen (SciGen Israel Ltd., produced in a new production facility located in Rehovot, Israel) contains three recombinant proteins of hepatitis B virus (HBV) envelope: small S, medium pre-S2, and large pre-S1 surface antigens. Sci-B-Vac-SciGen was supplied in a final volume of 1.2 ml vials
  Interventions: Biological: Sci-B-Vac-Lot B
- Engerix-B (Active Comparator): The single antigen HepB vaccine, Engerix-B (GSK), contains the small S recombinant protein. Engerix-B was supplied in 1.0 ml vials.
  Interventions: Biological: Engerix-B
- Sci-B-Vac-BTG (Experimental): The 3-antigen HepB vaccine, Sci-B-Vac-BTG (Bio-Technology General (BTG) Ltd., Rehovot, Israel.) contains three recombinant proteins of HBV viral envelope: small S, medium pre-S2, and large pre-S1 surface antigens. Sci-B-Vac-BTG was supplied in a final volume of 1.2 ml vials
  Interventions: Biological: Sci-B-Vac-Lot A

INTERVENTIONS:
Biological: Sci-B-Vac-Lot B — Sci-B-Vac Lot B -10 μg of HBsAg, intramuscular injection of 10 μg/ml
  Other Names: Sci-B-Vac; 3-antigen HepB Vaccine; Bio-Hep-B
  Arms: Sci-B-Vac-SciGen
Biological: Sci-B-Vac-Lot A — Sci-B-Vac Lot A - 10 μg of HBsAg, intramuscular injection of 10 μg/ml
  Other Names: Sci-B-Vac; 3-antigen HepB Vaccine; Bio-Hep-B
  Arms: Sci-B-Vac-BTG
Biological: Engerix-B — Engerix-B (hepatitis B vaccine (recombinant)) is indicated for active immunization against hepatitis B virus infection
  Arms: Engerix-B

SUMMARY:
This was a single-blind, 3-arm, comparative, controlled, randomized, study conducted at one site in Vietnam whose primary objective was to demonstrate clinical equivalence of the two production lots of Sci-B-Vac vaccine produced at two different facilities (OLD facility (Lot A) and NEW facility (Lot B) with respect to anti-hepatitis B-Surface (HBs) response. Secondary efficacy analysis was performed to demonstrate non-inferiority of seroprotection of each lot of Sci-B-Vac vaccine when compared to Engerix-B vaccine

DETAILED DESCRIPTION:
This was a single-blind, 3-arm, comparative, controlled, randomized, study conducted at one site in Vietnam. Following a screening period, healthy eligible subjects (n = 402) were enrolled and randomized to receive Sci-B-Vac (OLD facility (Lot A) and NEW facility (Lot B), or Engerix-B.

The study was conducted in two stages, approximately a year-and-a-half apart. In the first stage (Stage I) beginning in March 2006, Sci-B-Vac (Lot A) vaccine was compared to Engerix-B; and in the second stage (Stage II) beginning in November 2007, the Sci-B-Vac (Lot B) vaccine was compared to Engerix-B. The subjects assigned to the Engerix-B group were equally divided between the stages, 67 subjects in the Engerix-B group in Stages I and II, respectively, for a total of 134 subjects, such that the final number of randomized subjects in Stage 1 and Stage 2 across the Sci-B-Vac Lot A, Sci-B-Vac Lot B and Engerix-B was 1:1:1, respectively. Immunogenicity evaluations for Stage I data (Visits 5 and 6) were conducted together with Stage II data.

ELIGIBILITY:
Inclusion Criteria:

Healthy adults 18 to 45 years of age who were seronegative for HBsAg, anti-HBs, anti-Hepatitis B core antigen, HIV, and Hepatitis C Virus (HCV)

Exclusion Criteria:

* Evidence of alcoholism or drug abuse, history of HIV, or HCV
* Blood transfusions within the three months prior to inclusion in the study
* Uncontrolled hypertension and other cardiovascular diseases
* Chronic/concurrent administration (>14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. Inhaled and topical steroids were permitted
* History of anaphylaxis (including shock) or any significant allergy or atopy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 402 (Actual)
Dates: Start 2006-03-02 (Actual); Primary Completion 2008-12-31 (Actual); Study Completion 2008-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Do G Canh, MD, Principal Investigator — National Institute of Hygiene and Epidemiology (NIHE), Hanoi, Vietnam
Locations (1):
- National Institute of Hygiene and Epidemiology (NIHE), Hanoi, Vietnam

REFERENCES:
- [Derived] Diaz-Mitoma F, Popovic V, Spaans JN. Assessment of immunogenicity and safety across two manufacturing lots of a 3-antigen hepatitis B vaccine, Sci-B-Vac(R), compared with Engerix-B(R) in healthy Asian adults: A phase 3 randomized clinical trial. Vaccine. 2021 Jun 29;39(29):3892-3899. doi: 10.1016/j.vaccine.2021.05.067. Epub 2021 Jun 8. PMID 34116873

RESULTS

PARTICIPANT FLOW:
Groups:
- Sci-B-Vac-Lot B: The 3-antigen HepB vaccine, Sci-B-Vac-Lot B (SciGen Israel Ltd., New Facility) contains10 μg of HBsAg/preS1/S2 injected intramuscularly at 10 μg/ml
- Engerix-B: The single-antigenic HepB vaccine, Engerix-B (GSK), contains the small S recombinant protein indicated for active immunization against hepatitis B virus infection. Engerix-B was supplied in 1.0 ml vials.
- Sci-B-Vac-Lot A: The 3-antigen HepB vaccine, Sci-B-Vac-Lot A (Bio-Technology General (BTG) Ltd., Old Facility) contains10 μg of HBsAg/preS1/S2 injected intramuscularly at 10 μg/ml
Period: Stage I
Arm/Group | Sci-B-Vac-Lot B | Engerix-B | Sci-B-Vac-Lot A
Started | 0 | 67 | 134
Completed | 0 | 62 | 116
Not Completed | 0 | 5 | 18
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 5 | 10
Period: Stage II
Arm/Group | Sci-B-Vac-Lot B | Engerix-B | Sci-B-Vac-Lot A
Started | 134 | 67 | 0
Completed | 121 | 57 | 0
Not Completed | 13 | 10 | 0
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0
Not completed — Moved from study area | 8 | 5 | 0

BASELINE CHARACTERISTICS:
Population: Safety was evaluated in all study participants who received at least one vaccination and for whom there was safety information.
Groups:
- Engerix-B: The mono-antigenic HepB vaccine, Engerix-B (GSK), contains the small S recombinant protein indicated for active immunization against hepatitis B virus infection. Engerix-B was supplied in 1.0 ml vials.
- Sci-B-Vac-Lot A: The 3-antigen HepB vaccine, Sci-B-Vac-Lot A (Old Facility) contains10 μg of HBsAg/preS1/S2 injected intramuscularly at 10 μg/ml
- Total: Total of all reporting groups
Arm/Group | Sci-B-Vac-Lot B | Engerix-B | Sci-B-Vac-Lot A | Total
Number analyzed (Participants) | 131 | 133 | 134 | 398
Age, Categorical [Count of Participants; unit: Participants] — Population: Available Observations
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 131 | 133 | 134 | 398
    >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Available Observations
  years | 20.58 (1.577) | 20.48 (1.655) | 20.79 (2.392) | 20.62 (1.913)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Available Observations
  Participants
    Female | 94 | 89 | 89 | 272
    Male | 37 | 44 | 45 | 126
Region of Enrollment [Count of Participants; unit: Participants]
  Vietnam | 131 | 133 | 134 | 398
Ethnic Group [Count of Participants; unit: Participants]
  White/Caucasian | 0 | 0 | 0 | 0
  Black | 0 | 0 | 0 | 0
  Asian | 131 | 133 | 134 | 398
  Other | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 50.2 (5.9) | 50.2 (7.3) | 51.8 (6.0) | 50.8 (6.5)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 20.1 (1.5) | 20.0 (2.2) | 20.9 (1.9) | 20.3 (1.9)
Smoking status [Count of Participants; unit: Participants]
  Smoker | 3 | 6 | 1 | 10
  Non-smoker | 128 | 127 | 133 | 388

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Antibody Response (≥10 IU/Liter) to Hepatitis B Surface Antigens One Month After the Third Vaccination
Description: Percentage of participants with an antibody response to hepatitis B surface antigens (anti-HBs), defined as an anti-HBs titer ≥10 IU/liter, one month after the third vaccination (Day 210) in the According-to-Protocol (ATP) population.
Time Frame: Day 210
Population: The according-to-protocol (ATP) population included all participants who received the three vaccinations, the third vaccination measurement of anti-HBs titers, and had no major protocol violations.
Measure: Count of Participants; unit: Participants
Arm/Group | Sci-B-Vac-Lot B | Engerix-B | Sci-B-Vac-Lot A
Number analyzed (Participants) | 120 | 117 | 112
Participants | 120 | 115 | 109

2. Secondary Outcome: Percentage of Participants With an Anti-HBs Antibody Titer ≥10 IU/Liter at Days 180, 210 and 360.
Description: Percentage of participants with an anti-HBs antibody response, defined as an anti-HBs titer ≥10 IU/liter, just prior to the third vaccination (Day 180) and 1 month (Day 210) and 6 months (Day 360) after the third vaccination in the According-to-Protocol (ATP) population.
Time Frame: Days 180, 210, and 360
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sci-B-Vac-Lot B | Engerix-B | Sci-B-Vac-Lot A
Number analyzed (Participants) | 120 | 117 | 112
Participants
  Day 180 | 118 | 95 | 102
  Day 210 | 120 | 115 | 109
  Day 360: number analyzed (Participants) | 116 | 112 | 105
  Day 360 | 115 | 110 | 101

3. Secondary Outcome: Anti-HBs Geometric Mean Concentration (GMC)
Description: Geometric mean concentration (GMC) of anti-HBs antibody just prior to the third vaccination (Day 180) and 1 month (Day 210) and 6 months (Day 360) after the third vaccination in the According-to-Protocol (ATP) population.
Time Frame: Days 180, 210, and 360
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/Liter
Arm/Group | Sci-B-Vac-Lot B | Engerix-B | Sci-B-Vac-Lot A
Number analyzed (Participants) | 120 | 117 | 112
IU/Liter
  Day 180 | 328.64 [237.01 to 455.69] | 44.42 [31.90 to 61.85] | 147.30 [105.02 to 206.60]
  Day 210 | 12,158.94 [8666.37 to 17059.02] | 4,124.24 [2926.93 to 5811.33] | 3,587.30 [2526.67 to 5093.16]
  Day 360: number analyzed (Participants) | 116 | 112 | 105
  Day 360 | 3188.68 [2249.17 to 4520.63] | 991.07 [694.76 to 1413.77] | 1239.82 [859.07 to 1789.33]

4. Secondary Outcome: Percentage of Participants With an Anti-HBs Antibody Titer ≥100 IU/Liter at Days 180, 210 and 360.
Description: Percentage of participants with an anti-HBs antibody response, defined as an anti-HBs titer ≥100 IU/liter, just prior to the third vaccination (Day 180) and 1 month (Day 210) and 6 months (Day 360) after the third vaccination in the According-to-Protocol (ATP) population.
Time Frame: Days 180, 210 and 360
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sci-B-Vac-Lot B | Engerix-B | Sci-B-Vac-Lot A
Number analyzed (Participants) | 120 | 117 | 112
Participants
  Day 180 | 99 | 40 | 68
  Day 210 | 118 | 113 | 106
  Day 360: number analyzed (Participants) | 116 | 112 | 105
  Day 360 | 113 | 100 | 94

ADVERSE EVENTS:
Time Frame: Subjects were assessed for safety at baseline, during treatment (Day 30, Day 180) and during follow up (Day 210, Day 310).
Description: Adverse events (AEs) were reported throughout the study and were rated by the investigator for severity and causality. All serious AEs (SAEs) and fatalities were reported immediately. Local and systemic solicited adverse reactions were recorded after each vaccination on participant diary cards. AEs were rated by the investigators for severity and causality. All fatalities and SAE were reported to SciGen Ltd and Pharmacovigilance of Quintiles Asia Pacific, Singapore.
Arm/Group | Sci-B-Vac-Lot B | Engerix-B | Sci-B-Vac-Lot A
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/133 | 0/134
Serious Adverse Events (participants affected / at risk) | 1/131 | 4/133 | 3/134
Other Adverse Events (participants affected / at risk) | 63/131 | 26/133 | 83/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sci-B-Vac-Lot B (N=131) | Engerix-B (N=133) | Sci-B-Vac-Lot A (N=134)
schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
hepatitis B (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
gastritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sci-B-Vac-Lot B (N=131) | Engerix-B (N=133) | Sci-B-Vac-Lot A (N=134)
Injection site pain (General disorders) | 57 | 19 | 79
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 3 | 18
Fatigue (General disorders) | 10 | 6 | 14
Malaise (General disorders) | 3 | 4 | 12
Injection site pruritus (General disorders) | 4 | 3 | 7
Pyrexia (General disorders) | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 3
Dizziness (Cardiac disorders) | 1 | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes